CLINICAL TRIAL: NCT00003206
Title: A Phase II Trial of Carboplatin Plus Paclitaxel in the Treatment of Locally Recurrent or Metastatic Nasopharyngeal Carcinoma
Brief Title: Carboplatin and Paclitaxel in Treating Patients With Locally Recurrent or Metastatic Nasopharyngeal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066059; E-2397
Record Dates: First submitted 1999-11-01; First posted 2004-06-16 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Cancer
Keywords: stage IV nasopharyngeal cancer; recurrent nasopharyngeal cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Nasopharyngeal Neoplasms | interventions — Carboplatin; Paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of carboplatin and paclitaxel in treating patients with locally recurrent or metastatic nasopharyngeal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the response and toxicity of carboplatin in combination with paclitaxel in patients with locally recurrent or metastatic nasopharyngeal carcinoma.

OUTLINE: Patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes. This cycle is repeated every 3 weeks. Patients may receive 6-8 cycles of therapy in the absence of toxicity and disease progression. Patients are followed every 3 months for the first 2 years, every 6 months for the next 3 years, and yearly thereafter.

PROJECTED ACCRUAL: 30 eligible patients will be accrued in approximately 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed locally recurrent or metastatic nasopharyngeal carcinoma that is not curable with resection or radiation therapy Bidimensionally measurable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count greater than 1500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL Renal: Creatinine less than 3.0 mg/dL Other: No active infections Serum calcium within institutional normal range No history of hypercalcemia Prior malignancy other than nasopharyngeal carcinoma allowed No concurrent malignancy Not pregnant or lactating Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior biologic therapy allowed Chemotherapy: No prior chemotherapy for metastatic or recurrent disease Prior induction or adjuvant chemotherapy concurrent with radiation therapy allowed No prior treatment with paclitaxel Endocrine therapy: Not specified Radiotherapy: See Chemotherapy Surgery: Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10-06 (Actual); Primary Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A. Murphy, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (18):
- United States (17):
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Lakeside), Chicago, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - University of Rochester Cancer Center, Rochester, New York
  - Ireland Cancer Center, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt Cancer Center, Nashville, Tennessee
- Pretoria Academic Hospital, Pretoria, South Africa